CLINICAL TRIAL: NCT00004025
Title: Phase I/II Trial of the Safety, Immunogenicity, and Efficacy of Autologous Dendritic Cells Transduced With Adenoviruses Encoding the MART-1 and gp100 Melanoma Antigens Administered With or Without Low Dose Recombinant Interleukin-2 (rIL-2) in Patients With Stage IV Melanoma
Brief Title: Vaccine Therapy With or Without Interleukin-2 in Treating Patients With Stage III or Stage IV Melanoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Genzyme, a Sanofi Company (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067245; GENZ-ML98-0501; DFCI-98258
Record Dates: First submitted 1999-11-01; First posted 2003-10-29 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2002-07

CONDITIONS: Melanoma (Skin)
Keywords: stage III melanoma; stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — aldesleukin

INTERVENTIONS:
Biological: aldesleukin
Biological: dendritic cell-gp100-MART-1 antigen vaccine

SUMMARY:
RATIONALE: Vaccines made from a person's white blood cells combined with melanoma antigens may make the body build an immune response to tumor cells. Interleukin-2 may stimulate a person's white blood cells to kill melanoma cells. Combining vaccine therapy with interleukin-2 may be an effective treatment for stage III or stage IV melanoma.

PURPOSE: Phase I/II trial to study the effectiveness of vaccine therapy with or without interleukin-2 in treating patients who have stage III or stage IV melanoma that cannot be surgically removed.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the safety, dose-limiting toxicity, and maximum tolerated dose of autologous dendritic cells transduced with adenoviruses encoding the MART-1 and gp100 melanoma antigens with or without interleukin-2 in patients with stage III or IV melanoma. II. Evaluate the cellular response and efficacy of these regimens in this patient population.

OUTLINE: This is a dose-escalation study. Patients are sequentially assigned to one of three dose levels. Patients receive modified autologous dendritic cells subcutaneously on day 1 with or without interleukin-2 IV on days 4-19. Treatment continues every 21 days for a total of 6 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of modified dendritic cells with or without interleukin-2 until the maximum tolerated dose (MTD) for each regimen is reached. The MTD is defined as the dose below that at which 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: Approximately 24-36 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed stage III or IV metastatic melanoma Unresectable disease for which no other therapy exists Measurable or evaluable disease by clinical or radiographic evaluation Metastatic tumor tissue expressing both gp100 and MART-1 No uncontrolled or progressive CNS involvement

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-1 Life expectancy: Not specified Hematopoietic: WBC at least 3,000/mm3 Platelet count at least 100,000/mm3 No clinically significant hematologic disorder Hepatic: Bilirubin less than 2.0 mg/dL No clinically significant hepatic disease Hepatitis B surface antigen negative Renal: Creatinine less than 2.0 mg/dL No clinically significant renal disease Cardiovascular: No clinically significant cardiac disease Other: Not pregnant or nursing Fertile patients must use effective contraception Negative pregnancy test HIV-1 and HIV-2 negative HTLV-1 negative No significant psychiatric disorder that would prevent compliance No underlying condition that would preclude study therapy No autoimmune disease or other major immune system illness No active infection requiring parenteral antibiotic therapy

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior immunotherapy with vaccines directed at MART-1 or gp100 melanoma antigens Prior interleukin-2 or interferon therapy allowed Chemotherapy: At least 4 weeks since prior chemotherapy and recovered No concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy and recovered Surgery: At least 4 weeks since prior surgery (except study biopsies) and recovered Other: At least 4 weeks since prior experimental therapy and recovered At least 4 weeks since prior immunosuppressive drugs and recovered No other concurrent experimental therapy or anti-cancer drugs No concurrent immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 1999-03

CONTACTS AND LOCATIONS:
Overall Officials: Amy E. Bock, Study Chair — Genzyme, a Sanofi Company
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - U.S. Oncology, Houston, Texas